CLINICAL TRIAL: NCT03215069
Title: Empagliflozin and the Preservation of Beta-cell Function in Women with Recent Gestational Diabetes
Acronym: EMPA post-GDM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-0226-A
Record Dates: First submitted 2017-07-07; First posted 2017-07-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes, SGLT-2 inhibitor, empagliflozin
MeSH Terms: conditions — Diabetes, Gestational | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin 10 mg PO daily
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): Matched placebo PO daily
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Empagliflozin 10 mg PO daily
  Arms: Empagliflozin
Drug: Placebo oral capsule — Placebo PO daily
  Arms: Placebo

SUMMARY:
Double-blind, parallel arm, randomized controlled trial, in which non-lactating women with recent GDM who are between 6 to 36 months postpartum to be randomized to either empagliflozin 10 mg daily or matching placebo. The duration of treatment will be 48-weeks. Beta-cell function will be assessed by Insulin Secretion-Sensitivity Index-2 (ISSI-2), measured on oral glucose tolerance test (OGTT) at baseline, 24-weeks, 48-weeks, and after a 4-week washout.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM), defined as glucose intolerance of varying severity with first onset and recognition in pregnancy, identifies a population of women who are at high risk for the future development of type 2 diabetes (T2DM). This risk of T2DM is mediated by the progressive deterioration of insulin secretion by the pancreatic beta-cells in the years after delivery, a pathologic process that current anti-diabetic therapies have not been shown to modify. Importantly, since very mild glycemia has deleterious but reversible effects on insulin secretion ("glucotoxicity"), the beta-cell dysfunction of women with recent GDM should have a prominent reversible component that potentially could be mitigated through the elimination of glucotoxicity. In this context, the sodium glucose co-transporter-2 (SGLT-2) inhibitor empagliflozin is a novel anti-diabetic therapy that specifically alleviates glucotoxicity and thus may be able to preserve beta-cell function. Coupled with its capacity to induce weight loss with low risk of hypoglycemia, empagliflozin could be an ideal therapy for diabetes prevention in women with recent GDM. Specifically, by eliminating glucotoxicity, SGLT-2 inhibition could enable the preservation of beta-cell function and thereby prevent the development of incident T2DM in this high-risk population. Thus, a double-blind, parallel arm, randomized controlled trial, in which non-lactating women with recent GDM who are between 6 to 36 months postpartum to be randomized to either empagliflozin 10 mg daily or matching placebo is proposed. The duration of treatment will be 48-weeks. Beta-cell function will be assessed by Insulin Secretion-Sensitivity Index-2 (ISSI-2), measured on oral glucose tolerance test (OGTT) at baseline, 24-weeks, 48-weeks, and after a 4-week washout.

ELIGIBILITY:
Inclusion Criteria:

* Women with recent gestational diabetes who are between 6-36 months postpartum inclusive and no longer breastfeeding
* Age 20 - 50 years inclusive
* Negative pregnancy test at recruitment

Exclusion Criteria:

* Current breastfeeding
* Current diabetes or treatment with any anti-diabetic medication
* Involvement in any other clinical study requiring drug therapy
* Hypersensitivity to empagliflozin or the formulations of this product
* Any history of diabetic ketoacidosis
* History of recurrent urinary infection (i.e. more than 2 episodes over the past year).
* Renal dysfunction as evidenced by estimated glomerular filtration rate < 45 ml/min by Modification of Diet in Renal Disease (MDRD) formula
* Hepatic disease considered to be clinically significant (includes jaundice, chronic hepatitis, or previous liver transplant) or transaminases >2.5X the upper limit of normal
* Malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy within the previous 5 years (with the exception of basal cell skin cancer)
* Pregnancy or unwillingness to use reliable contraception. Women should not be planning pregnancy for the duration of the study or the first 3 months after the study. Reliable contraception includes the following: birth control pill, intra-uterine device, abstinence, tubal ligation, partner vasectomy, or condoms with spermicide.
* Any other factor likely to limit adherence to the study, in the opinion of the investigators

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with history of gestational diabetes
Enrollment: 91 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted ISSI-2 at 48-weeks | 48-weeks
  The primary outcome will be measured by ISSI-2. ISSI-2 is a validated OGTT-derived measure of beta-cell function analogous to the disposition index obtained from the intravenous glucose tolerance test. ISSI-2 is defined as the product of (i) insulin secretion measured by the ratio of the area-under-the-insulin-curve (AUCins) to the area-under-the-glucose curve (AUCgluc) and (ii) insulin sensitivity measured by the Matsuda index.

SECONDARY OUTCOMES:
Glucose tolerance status at 48-weeks | 48-weeks
  Prevalence of dysglycemia on the OGTT at this visit.

OTHER OUTCOMES:
Baseline-adjusted ΔISR0-120/Δgluc0-120 × Matsuda index at 48 weeks | 48-weeks
  and insulinogenic index/HOMA-IR.
Baseline-adjusted insulinogenic index/HOMA-IR at 48-weeks | 48-weeks
  Beta-cell function assessed by ΔISR0-120/Δgluc0-120 × Matsuda index at 48-weeks
Body mass index at 48-weeks | 48-weeks
Insulin sensitivity at 48 weeks. | 48-weeks
  Insulin sensitivity will be measured by Matsuda index on OGTT
Central abdominal fat mass at 48 weeks | 48-weeks
  Central abdominal fat mass will be measured by DXA assessment at L2-L4
Quality of life at 48 weeks | 48-weeks
  Quality of life will be assessed annually by the Medical Outcomes Study 36-item Short-Form Health Survey (SF-36).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline kramer, MD PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Leadership Sinai Centre foe Diabetes - Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murugavel S, Retnakaran R, Feig DS, Zinman B, Kramer CK. Empagliflozin for the preservation of beta-cell function in women with recent gestational diabetes: A randomized placebo-controlled trial. Diabetes Obes Metab. 2025 Dec;27(12):7408-7415. doi: 10.1111/dom.70146. Epub 2025 Sep 18. PMID 40964955